CLINICAL TRIAL: NCT06560827
Title: A Single-arm, Open-label, Multicenter, Phase Ib Clinical Trial to Evaluate the Safety and Efficacy of CT011 Autologous CAR-T Cells in Patients With Hepatocellular Carcinoma at Risk of Recurrence After Surgical Resection
Brief Title: CT011 Autologous CAR-T Cells in Patients With Hepatocellular Carcinoma at Risk of Recurrence After Surgical Resection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT011-HCC-03
Record Dates: First submitted 2024-07-25; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: HCC
Keywords: IIIa; GPC3; HCC; CT011

STUDY DESIGN:
Intervention Model Description: It is planned to enroll approximately 30 participants to receive CT011 infusion.
  During the trial, the sample size may be appropriately adjusted as assessed by the sponsor and the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT011 CAR-GPC3 T Cells Injection (Experimental): This trial is a single-arm, open-label, exploratory trial, and no statistical hypothesis is made for sample size estimation. It is planned to enroll approximately 30 participants to receive CT011 infusion.
  Interventions: Biological: CT011 CAR-GPC3 T Cells Injection

INTERVENTIONS:
Biological: CT011 CAR-GPC3 T Cells Injection — The dose selection for this trial was mainly based on the preliminary safety and efficacy results of CT011-HCC-01 trial in subjects with advanced HCC, in which 3 and 5 subjects in the 2.5 × 108 cell and 5.0 × 108 cell dose groups, respectively, completed a single infusion of CT011. The results showed that the two dose groups of CT011 were generally well tolerated in HCC subjects who failed to standard treatment, with controllable safety, and showed preliminary anti-tumor efficacy.

SUMMARY:
A Single-arm, Open-label, Multicenter, Phase Ib Clinical Trial to Evaluate the Safety and Efficacy of CT011 Autologous CAR-T Cells in Patients with Hepatocellular Carcinoma at Risk of Recurrence after Surgical Resection.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, exploratory phase Ib clinical trial to evaluate the safety, efficacy, and cellular kinetics of CT011 CAR-GPC3 T cells (referred to as CT011) in participants with CNLC stage IIIa, GPC3-positive HCC at risk of recurrence after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial, participants must meet all of the following criteria:

1. Volunteer to participate in the clinical trial; fully understand and are informed of this trial and sign the informed consent form; Willing to follow and able to complete all trial procedures;
2. Age 18-75 years, inclusive, male or female;
3. Initially diagnosed with CNLC stage IIIa HCC with any of the following vascular tumor thrombi and absence of atrial tumor thrombi on preoperative imaging:

   * Portal vein tumor thrombus (PVTT);
   * Hepatic vein tumor thrombus (HVTT);
   * Inferior vena cava tumor thrombus (IVCTT);
4. Has undergone surgical resection:

   * Pathological evaluation of surgical resection specimen with negative margins;
   * Preoperative conversion/neoadjuvant therapy and/or postoperative therapy are allowed;
5. The participant has recovered from liver resection and postoperative progressive increase in AFP level(including: a. AFP increase of at least 20% in any 3 months after surgery; or b. AFP increase of ≥ 10% in any 2 consecutive tests after surgery) with a potential tendency to recurrence as assessed by the investigator.
6. Tumor tissue samples positive for GPC3 by immunohistochemistry (IHC) (staining intensity ≥ 1 +, percentage of stained tumor cells ≥ 10%);
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (within 7 days prior to apheresis);
8. Child-Pugh score ≤ 7 points (within 7 days prior to apheresis);
9. Estimated survival > 12 weeks;
10. Adequate venous access for apheresis;
11. Laboratory test results within 7 days prior to apheresis should meet the following criteria (if the laboratory test results do not meet the following criteria, a repeat test within 1 week is allowed; if the laboratory test results still do not meet the criteria, it will be considered a screening failure):

    * Hematology (without transfusion, platelet transfusion, colony-stimulating factor and other supportive treatment within 7 days before detection, except recombinant human erythropoietin): neutrophil count (ANC) ≥ 1.5 × 109/L, lymphocyte count (LY) ≥ 0.5 × 109/L, platelet count (PLT) ≥ 75 × 109/L, hemoglobin (Hb) ≥ 9.0 g/dL; The results of hematology within 24 hours before apheresis shall also meet this standard;
    * Blood chemistry: serum creatinine ≤ 1. 5 × upper limit of normal (ULN), endogenous creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault formula), alanine aminotransferase (ALT) ≤ 5×ULN, aspartate aminotransferase (AST) ≤ 5 × ULN, alkaline phosphatase (ALP) ≤ 5 × ULN, total bilirubin (TBil) ≤ 3 × ULN, serum albumin (ALB) ≥ 28 g/L, and serum lipase and amylase ≤ 2 × ULN;
    * Prothrombin time (PT) prolongation ≤ 4 s;
12. Female participants of childbearing potential must have a negative serum pregnancy test at screening and agree to remain abstinent or use highly effective and reliable contraception (< 1% failure rate per year) during the treatment period and for at least 1 year after the last dose of trial treatment, during which time they must not donate eggs:

    * Women of childbearing potential are defined as women who have not reached post-menarche but have not reached a post-menopausal state (no menses for ≥ 12 consecutive months, with no cause other than menopause) and who have not been permanently infertile due to surgery (removal of ovaries, fallopian tubes, and/or uterus) or other reasons (e.g. M ü llerian agenesis, etc.) as determined by the investigator;
    * Contraceptive methods with an annual failure rate of < 1% include: bilateral tubal ligation, male sterilization, approved hormonal contraceptives, hormone-releasing intrauterine devices, copper-containing intrauterine devices; Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation rhythm methods) and withdrawal are not adequate methods of contraception.
13. Male participants who are sexually active with a female of childbearing potential, who have not had a vasectomy, must agree to remain abstinent or to use contraception (e.g., condoms in combination with other contraceptive measures to achieve an annual failure rate of < 1%, see inclusion criterion # 12) during the treatment period and for 1 year after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

Participants were not included in the trial if they met any of the following criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed hepatocellular-cholangiocarcinoma;
2. Intrahepatic recurrence or extrahepatic metastasis, or residual hepatocellular carcinoma detected before apheresis (imaging evidence according to RECIST v1.1);
3. More than 2 years since surgical resection;
4. Pregnant or lactating females;
5. Positive test results for any of the following: human immunodeficiency virus (HIV) antibody, Treponema pallidum antibody, hepatitis C virus (HCV) ribonucleic acid (RNA), hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive and hepatitis B virus deoxyribonucleic acid [HBV DNA] ≥ 1000 IU/mL (HBsAg-positive or HBcAb-positive participants must receive antiviral therapy), cytomegalovirus (CMV) DNA, Epstein-Barr virus (EBV) DNA;
6. Any uncontrolled active infection, including but not limited to active tuberculosis, infectious diseases requiring systemic treatment, etc.; Patients who use drugs to prevent infection can be enrolled at the discretion of the investigator;
7. Subjects with clinically significant abnormal thyroid function (free triiodothyronine [FT3], free thyroxine [FT4] and serum thyroid stimulating hormone [TSH] for serum thyroid hormones, and total thyroxine [TT4] and total triiodothyronine [TT3] for serum thyroid hormones if necessary) judged by the investigator and not suitable for entry into the trial after assessment; Patients with stable thyroid function after treatment can be considered for inclusion;
8. Previous or current hepatic encephalopathy;
9. Presence of clinically significant massive abdominal/pleural effusion, defined as: positive signs of pleural/peritoneal effusion on physical examination or pleural/peritoneal effusion requiring intervention (e.g., paracentesis or drug therapy) for control;
10. Toxicities caused by previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 ≤ Grade 1, except for alopecia, pigmentation, other laboratory abnormalities that do not affect the tolerability of the participants as judged by the investigator;
11. Received anti-tumor treatment for the disease under study within 2 weeks prior to apheresis, including but not limited to surgery, systemic drug therapy (or within 5 half-lives of the drug, whichever is shorter), radiotherapy, interventional therapy, etc.;
12. Received immunotherapy including anti-PD-1/PD-L1, anti-CTLA-4, or any other investigational therapy within 4 weeks (or within 5 half-lives of the drug, whichever is shorter) prior to apheresis;
13. Previously received any cell therapy (including CAR-T cells, TCR-T cells, TILs, etc.);
14. Received systemic glucocorticoid therapy within 7 days prior to apheresis; Patients with recent or current use of inhaled or topical corticosteroids and physiologic dose replacement therapy may be enrolled;
15. Vaccination with live or live attenuated vaccines within 4 weeks prior to apheresis or planned during the trial;
16. Known active autoimmune disease, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, autoimmune hepatitis, interstitial lung disease, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, multiple sclerosis, glomerulonephritis, etc.; Or other participants who require chronic use of immunosuppressive therapy;
17. Participants with a history of organ transplantation, allogeneic hematopoietic stem cell transplantation or awaiting organ transplantation;
18. Previous allergies to immunotherapy, tocilizumab, cyclophosphamide or fludarabine and other related drugs, previous history of severe allergies, or known allergies to components of CT011 cell infusion preparation (such as albumin or dimethyl sulfoxide, etc.);
19. Presence of central nervous system metastasis or related symptoms, or clinically significant central nervous system disease or abnormal neurological examination results or psychiatric disease;
20. Need for long-term anticoagulation/thrombolysis/antiplatelet therapy (such as warfarin, heparin, rivaroxaban, aspirin, dipyridamole, clopidogrel, etc.); Patients receiving prophylactic anticoagulation to maintain patency of venous access devices may be included in this trial;
21. Major surgical procedure or significant trauma within 4 weeks prior to apheresis, or anticipation of the need for major surgery during the trial;
22. Pre-apheresis oxygen saturation ≤ 95% (under room air, the finger pulse oxygen test is accepted);
23. Any other disease, metabolic disorder, sign, or test result that contraindicates the use of the trial drug, affects the interpretation of the results, or places the participant at high risk of treatment complications, which, as assessed by the investigator, would not be appropriate for participation in the trial, including but not limited to: poorly controlled diabetes mellitus (treated glycosylated hemoglobin [HbA1c] > 8%), poorly controlled hypertension (blood pressure > 160 mmHg/100 mmHg), hypotension requiring vasopressor medication, uncontrolled congestive heart failure (New York Heart Association [NYHA] Class III-IV), Left ventricular ejection fraction [LVEF] < 50%, myocardial infarction within the past 6 months, arrhythmia not well controlled by drug therapy, unstable angina pectoris, or other serious heart disease, pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease or clinically significant pulmonary function test abnormality as judged by the investigator; Presence of currently gastrointestinal obstruction or active/unstable gastrointestinal ulcer, gastrointestinal bleeding within the past 3 months or with bleeding risk (e.g., esophageal and gastric varices caused by portal hypertension or bleeding tendency; patients with liver cirrhosis are recommended to undergo additional gastroscopy during the screening period according to the judgment of the investigator to determine the condition of varices); The participant is in a severe inflammatory state overall (e.g., increased neutrophil count and/or C-reactive protein, fever ≥ 38 ℃ unrelated to the underlying disease);
24. Presence of other incurable malignancies within the past 5 years or at the same time, except for appropriately treated cervical carcinoma in situ, skin basal cell carcinoma and other malignancies with very low risk of metastasis/death;
25. Inability or unwillingness of the participant to comply with the requirements of the trial protocol as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAE) | Up to 12 months
  According to the two-level classification of System Organ Classification (SOC) and Preferred Term, calculate the number and incidence of each type of AE separately; List and describe the severity of AE and its relationship with experimental treatment.
Incidence and severity of treatment-related adverse events (TRAE) | Up to 12 months
  List the AE related to the experimental treatment separately, and calculate the number and incidence of adverse events (TRAEs) related to the experimental treatment.
Incidence and severity of adverse events of special interest (AESI) | Up to 12 months
  Regardless of the causal relationship, the following events occurring after CAR-T cell infusion until 12 months after the last infusion are considered AESI: any ≥ grade 3 CRS; ≥ Level 3 HLH; Any ICANS level ≥ 3; Any grade ≥ 2 infusion related reaction (IRR); Any grade 3 or higher allergic reactions, etc. Evaluate the incidence and rate of AESI.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | Up to 12 months
  The time from the first infusion (D0) to the occurrence of intrahepatic recurrence/extrahepatic metastasis or death from any cause, whichever occurs first.
W24, W48, and W72 RFS rates | Up to 12 months
  The proportion of participants who survived and did not experience intrahepatic recurrence/extrahepatic metastasis at W24, W48, and W72 after the first infusion (D0).
Time to recurrence (TTR) | Up to 12 months
  The time from the first infusion (D0) to the first recording of intrahepatic recurrence and/or extrahepatic metastasis (whichever occurs first).
Time to intrahepatic recurrence (TT-IHR) | Up to 12 months
  The time from the first infusion (D0) to the first recording of intrahepatic recurrence.
Time to extrahepatic spread (TT-EHS) | Up to 12 months
  The time from the first infusion (D0) to the first recording of extrahepatic spread.
Postoperative recurrence free survival (RFS2) | Up to 12 months
  The time from liver resection surgery to the occurrence of intrahepatic recurrence/extrahepatic metastasis or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 12 months
  The time from the first infusion (D0) to the participant's death from any cause.
OS rates of W24, W48, and W72 | Up to 12 months
  the proportion of participants who survived W24, W48, and W72 after the first infusion (D0).
AFP control rate (ACR) of W24, W48, and W72 | Up to 12 months
  The proportion of participants whose AFP levels reached remission, decrease, and stability at W24, W48, and W72 after the first infusion (D0).
To evaluate the cellular metabolic kinetics of CT011 | Up to 12 months
  Time to peak expansion (Tmax)
To evaluate the cellular metabolic kinetics of CT011 | Up to 12 months
  peak expansion (Cmax)
To evaluate the cellular metabolic kinetics of CT011 | Up to 12 months
  area under the curve (AUC)
To evaluate the cellular metabolic kinetics of CT011 | Up to 12 months
  continuous survival time (Tlast) of CT011 cells after infusion
To evaluate the immunogenicity of CT011 | Up to 12 months
  Positive rate of anti-drug antibodies (ADA) after CT011 cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jia fan, Study Director — Fudan University
Locations (15):
- China (15):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Hunan Provincial People's Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing university ca cer hospital, Chongqing
  - Mengchao hepatobiliary hospital of fujian medical university, Fuzhou
  - Sun Yat-sen University Cancer Center, Guanzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The second affiliated hospital zhejiang university school of medicine, Hangzhou
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - The first hospital of china medical university, Shenyang
  - Tianjin medical university cancer hospital, Tianjin
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou